CLINICAL TRIAL: NCT06868082
Title: A Phase 1, Open-Label Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Two Formulations of Subcutaneously Administered Solrikitug in Healthy Japanese and Non-Japanese Participants
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics of Solrikitug in Healthy Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uniquity One (UNI) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSI-8226-102
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A Solrikitug (Experimental)
  Interventions: Biological: Solrikitug
- Cohort B Solrikitug (Experimental)
  Interventions: Biological: Solrikitug
- Cohort C Solrikitug (Experimental)
  Interventions: Biological: Solrikitug

INTERVENTIONS:
Biological: Solrikitug — Solrikitug Formulation 1
  Arms: Cohort A Solrikitug
Biological: Solrikitug — Solrikitug Formulation 2
  Arms: Cohort B Solrikitug; Cohort C Solrikitug

SUMMARY:
A Phase 1, Open-Label Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Two Formulations of Subcutaneously Administered Solrikitug in Healthy Japanese and non-Japanese Participants

ELIGIBILITY:
Inclusion Criteria:

* At the time of initial screening, in general good health (age 18 to 55 years);
* Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring
* Participant must agree to use contraception during the treatment period and until follow-up
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions of the study

Exclusion Criteria:

* Pregnancy or breastfeeding during the study
* Chronic infection
* Treatment with prohibited medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 165 days
  Treatment-Emergent Adverse Events according to Common Terminology Criteria for Adverse Events (CTCAE) V4.0

SECONDARY OUTCOMES:
Serum concentration of solrikitug | 112 days
  Pharmacokinetics (PK) of solrikitug in healthy participants
Concentration of Immunogenicity | 112 days
  Immunogenicity profile of solrikitug in healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lee, MD, Study Chair — Uniquity One
Locations (1):
- Research Site, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol